CLINICAL TRIAL: NCT07336732
Title: A Phase II, Open-label, , Multicenter Study Evaluating the Efficacy and Safety of Andamertinib in Patients With Previously Untreated, Locally Advanced or Metastatic Non-squamous Non-Small Cell Lung Cancer Harboring EGFR PACC or EGFR L861Q Mutations.
Brief Title: Andamertinib as First-line Treatment for NSCLC With EGFR PACC or EGFR L861Q Mutation
Acronym: KANNON-5
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLB1004-II/III-01
Record Dates: First submitted 2025-12-18; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cance; EGFR; PACC; L861Q; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLB1004 given alone as monotherapy (Experimental): PLB1004 is a capsule in the form of 80mg and 40mg
  Interventions: Drug: PLB1004

INTERVENTIONS:
Drug: PLB1004 — PLB1004 is a capsule in the form of 80mg and 40mg

SUMMARY:
This study is an open-label, multicenter phase IIclinical trial designed to evaluate the efficacy, safety, and tolerability of Andamertinib (phase II) in previously untreated participants with locally advanced or metastatic non-squamous NSCLC harboring EGFR PACC mutations or EGFR L861Q mutations.

DETAILED DESCRIPTION:
This a three-stage study consist a Screening Phase (Day -28 to -1), a Treatment Phase (until treatment discontinuation), and a Follow-up Phase (including end of treatment visit (EOT),end of study visit(EOS), safety follow-up and survival follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of ICF signing.
2. Histologically or cytologically confirmed, unresectable locally advanced (Stage IIIB or IIIC) or metastatic (Stage IV) non-squamous non-small cell lung cancer (NSCLC).
3. Confirmed presence of EGFR PACC mutation or EGFR L861Q mutation.
4. No prior systemic therapy for locally advanced or metastatic NSCLC.
5. At least one measurable lesion as defined by RECIST v1.1.
6. ECOG PS ≤1.
7. Life expectancy≥12 weeks.
8. Adequate organ function confirmed within 7 days prior to the first dose of study treatment
9. Female participants must use adequate contraceptive measures during study participation and for 90 days after the last dose of study treatment and must not be breastfeeding; female subjects not of childbearing potential must meet at least one of the following criteria at screening: Postmenopausal status; Documentation of irreversible surgical sterilization.
10. Non-sterilized males: Abstinence or contraception use; No sperm donation.
11. Willing and able to provide signed ICF and to comply with all requirements and restrictions listed in the ICF and this study protocol.

Exclusion Criteria:

1. Presence of specific genetic alterations for which approved targeted therapies are available.
2. Recent participation (within 28 days) in another interventional clinical trial.
3. Major surgery within 28 days prior to study entry or planned during the study period.
4. Recent use of anti-tumor traditional proprietary medicine or local anti-tumor therapy.
5. Need for specific concomitant medications (e.g., metformin) that cannot be paused during the study.
6. History of another active malignancy within the past 5 years (except for specific cured cancers).
7. Toxicities from prior therapy have not recovered to acceptable levels.
8. Presence of symptomatic or uncontrolled brain metastases, carcinomatous meningitis, or spinal cord compression.
9. Symptomatic and uncontrolled third-space fluid accumulations (e.g., pleural effusion, ascites).
10. Severe cardiovascular/cerebrovascular disease or risk factors (e.g., heart failure, history of myocardial infarction, QT prolongation, uncontrolled hypertension, etc.).
11. History or presence of interstitial lung disease, or drug/radiation-related pneumonitis.
12. Active autoimmune or inflammatory diseases.
13. Active, uncontrolled infection (including HBV, HCV, HIV, syphilis, tuberculosis, etc.).
14. Gastrointestinal disorders or surgery affecting drug ingestion or absorption.
15. Active keratitis or ulcerative keratitis.
16. History of hypersensitivity to the study drug, its analogs, or chemotherapy drugs (pemetrexed/platinum agents).
17. Recent administration (within 30 days) of a live attenuated vaccine.
18. Psychiatric disorders or substance abuse potentially affecting compliance.
19. Any other condition deemed by the investigator as unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | Up to 3 years
  In phase II，Incidence of Treatment-Emergent Adverse Events (TEAEs)
RP3D | Up to 3 years
  In phase II, choose the RP3D per gained safety and efficacy data

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 3 years
  To evaluate the Overall Response Rate (ORR) which is defined by investigator as the proportion of subjects with confirmed best overall response of complete response or partial response per RECIST v1.1
Duration of Response(DOR) | up to 3 years
  DOR is defined as the time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes frst
Disease Control Rate(DCR) | up to 3 years
  The percentage of tumor patients achieving complete remission (CR), partial remission (PR), or stable disease (SD) following treatment, relative to the total number of evaluable subjects
Progression-Free Survival(PFS) | up to 3 years
  PFS is defined as the time from the date the first dose until the date of objective disease progression or death by cause whichever comes first, based on investigator review according to RECIST v1.1
6-month Progression-Free Survival Rate | up to 3 years
  The proportion of subjects who did not experience disease progression or death within 6 months after receiving treatment.
6-month Overall Survival Rate | up to 3 years
  The proportion of subjects who did not experience death within 6 months after receiving treatment.
Assess the PK characteristics of Andamertinib | On cycle1of day 1and cycle3of day1, samples were collected within 2 hours prior to dosing and 4 hours post-dosing,On Day 1of Cycle 2, Cycle 5, Cycle 7, and all subsequent odd-numbered cycles collected within 2hours prior to dosing(each cycle is 21days)
  Plasma concentration of Andamertinib